CLINICAL TRIAL: NCT01418456
Title: A Prospective Single Blind Randomised Controlled Study to Compare the Outcomes of Patients With Diabetes and Clinically Non-infected Neuro-ischaemic and Neuropathic Foot Ulcers Treated With and Without Oral Antibiotics.
Brief Title: Outcomes of Non-infected Diabetic Foot Ulcers With/Without Antibiotics
Acronym: KADFUT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Professor Mike Edmonds, King's College Hospital NHS Foundation Trust
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KADFUT; 2010-022518-16 (EudraCT Number)
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes; Foot Ulcers; Infection
Keywords: diabetes; antibiotics; clean foot ulcers
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Infections | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Antibiotic Group (Experimental): Patients in the antibiotic group will remain on antibiotics until their foot ulcer heals or up to 20 weeks
  Interventions: Drug: antibiotics
- Non antibiotic group (No Intervention)

INTERVENTIONS:
Drug: antibiotics — A variety of antibiotics may be used, according to microbiology results, for up to 20 weeks
  Arms: Active Antibiotic Group

SUMMARY:
The overall objective is to investigate whether antibiotics in the treatment of clinically clean neuropathic and ischaemic ulcers in diabetic foot patients could reduce the incidence of infection and therefore lead to improved outcomes This is a single centre study in which patients with either type 1 or 2 diabetes mellitus, who consecutively present to the Diabetic Foot Clinic [DFC] with clean neuropathic (NU) or ischaemic (IU) diabetic foot ulcer without clinical signs of infection will be invited to take part and will express their willingness to take part in the study by signing a consent form.

* All patients will be treated and followed up in the DFC at King's College Hospital. Patients will be randomised into two groups: an antibiotic group and a control group.
* The antibiotic group will receive standard treatment along with antibiotics.
* The control group will have standard treatment alone.
* Patients from both groups will be reviewed at weekly intervals for a period of 20 weeks.
* Patients will be removed from the study if they develop clinical signs of infection or if their ulcer heals prior to 20 weeks but will be followed up via routine practice for eventual outcomes

DETAILED DESCRIPTION:
Trail Procedures Visit 0 Screening, Randomisation and Initial Treatment;

1. The researcher will assign a screening number.
2. Medical history and demographics will be recorded.
3. Physical examination including height and weight will be performed.
4. Vital signs (body temperature, pulse and blood pressure) will be recorded.
5. Random capillary blood glucose will be measured.
6. Blood investigations as per routine clinical practice in the Diabetic Foot Clinic will be carried out including:

   Calcium and Phosphate Renal and liver function Glycated haemoglobin C- Reactive Protein (CRP) Full blood cell count Erythrocyte sedimentation rate Blood glucose Blood will also be taken for high sensitivity C-reactive protein, and procalcitonin levels as inflammatory markers. (Samples will be stored in a -80 deg C freezer, to be analysed at a later date)
7. A urine test for Beta human chorionic gonadotropin test for women of childbearing potential will be carried out
8. The foot ulcer will then be debrided of callous and any macerated tissue and details of the ulcer will be recorded as follows;
9. Ulcer characteristics and presence of signs of infection (redness, swelling, pain, malodour, purulent discharge) .
10. In order to enter the study, the patient will need to have a clinically non- infected ulcer.

    If patients have more than one ulcer, each ulcer should have no clinical signs of infection and the largest foot ulcer will be recorded as the target ulcer and will be monitored in the study. (The remaining ulcers will be treated according to standard clinical practice.)

    At this stage inclusion/ exclusion criteria will be reviewed and if satisfied, the patient will be admitted to the study.
11. The circumference of the ulcer selected for the study will be marked out using sterile graph paper and a marker pen.
12. A digital photograph will be taken. The patient will be asked to sign a consent form for this as part of King's College Hospital NHS Trust policy.
13. A tissue sample( ulcer biopsy) will be sent for culture and sensitivity
14. The foot ulcer will then be cleansed with normal saline. A sterile non adherent dressing along with a surgipad dressing will be applied to the foot ulcer. If appropriate the patient's usual carers can be shown the dressings to be used and be given training to ensure correct application of the dressings between visits to the clinic. Dressing changes should occur according to the amount of exudate discharging from the ulcer, ie. every day, every second, third day or three times a week. Patients will be advised to keep their ulcer dressings dry.

    VASCULAR ASSESSMENT
15. Palpation of pedal pulses namely dorsalis pedis and posterior tibial will be carried out. Ulcers occurring on the foot with impalpable pedal pulses will be defined as ischaemic ulcers.
16. If pulses are impalpable, ankle- brachial pressure index and transcutaneous oxygen (TcPo2) measurements will be performed and recorded. Patients will be reviewed by the vascular team together with their vascular studies. The vascular consultant, diabetes consultant and the patient will make a decision regarding any vascular intervention such as angioplasty or bypass or to continue with conservative management.
17. Patients who have ischaemic feet will have their TcPo2 monitored on a once monthly basis. If there is any deterioration in their blood supply they will be seen by the vascular team to consider vascular intervention with either by-pass or angioplasty or continue with monitoring.
18. A scotch cast boot (SCB) to optimise offloading for the ischaemic ulcer, will be manufactured for patients with impalpable pedal pulses as per standard clinical practice.

    NEUROLOGICAL ASSESSMENT
19. Peripheral sensation testing will be carried out using a neurothesiometer to determine vibration perception threshold on the apex of the toe of the foot with the ulcer. A 10g nylon monofilament will be applied to the plantar surface of the 1st toe, and to the plantar surface of the 1st ,3rd and 5th metatarsal heads and heel. Patients will be deemed to have neuropathy if the vibration perception threshold is abnormal or the filament cannot be felt on the plantar surface at any of the sites.

    Ulcers occurring on the foot with abnormal vibration perception or 10g filament testing will be defined as neuropathic ulcers.
20. A removable total contact cast (RTCC) to optimise offloading in the neuropathic ulcer, will be manufactured as per standard clinical practice.
21. All patients will be asked to complete:

    Quality of life questionnaire SF-36 EuroQol-5 questionnaire (EQ-5D)
22. All patients in the trial will be given emergency contact details.

Randomisation

* Patients will be randomised to one of two groups
* The antibiotic group
* The standard treatment only group

Antibiotics will be dispensed from the hospital pharmacy. Patients will be advised that there will always be two teams of health care professionals monitoring them: the blinded team, which is the team who do not know which treatment group the patient has been assigned, and the un blinded team, which is the team who do know what treatment group to which the patient has been assigned .The patient will be asked not to inform the blinded team as to which group they belong.

Visits 1-19

The unblinded team will always see the patient first.

Adverse events will be noted and assessed Adherence to treatment will be assessed and recorded Details of the resources that have been used by the patient for treatment of their ulcer will be recorded in order to carry out a health economic evaluation.

1. Vital signs will be recorded (body temperature, pulse and blood pressure).
2. Random capillary blood glucose will be measured.
3. Patients with ischaemic ulcers will have their TcPO2 measured at four weekly intervals weeks 4,8,12,16 and 20.

   The blinded team will carry out the following assessments;
4. Ulcer characteristics (size, depth, site).
5. Presence of clinical signs of infection such as; redness, swelling, pain, malodour, purulent discharge.
6. A tissue specimen from the ulcer bed will be sent for culture and sensitivity, at week 4,8,12,16 and 20. An ulcer swab will be taken at all other visits.
7. A digital photograph will be taken
8. The ulcer circumference will be marked out using sterile graph paper and a marker pen.
9. The SCB or RTCC will be checked with patient.
10. The ulcer will be cleansed using normal saline, a standard non adherent dressing and a surgipad dressing held in place with a bandage will be applied to the ulcer.
11. The ulcer will be deemed infected or non- infected.
12. The blinded team will inform the unblinded team whether the ulcer is healed ; if it is not healed, whether it is infected or non infected, using the Infectious Disease Society of America/International Working Group on the Diabetic Foot Guidelines (IDSA-IWGDF) criteria for infection. This will be confirmed by two members of the blinded team If the ulcer is deemed to be clinically non-infected, and patient is to continue in the study, antibiotics will be rationalised by the unblinded team according to culture and sensitivity results from the ulcer swab/biopsy. An appropriate clinical trial prescription will be written.
13. Emergency contact details will be checked with the patient.
14. Patients will be followed up to 20 weeks. The patient will be withdrawn from the study before the 20 weeks has elapsed if a foot ulcer has developed clinical signs of infection or the ulcer has healed or the patient has developed side effects necessitating the patient to stop antibiotic therapy for more than 72 hours or is withdrawn by the Investigator for any other reason.
15. If the patient is withdrawn early termination procedures will be completed (as per visit 20 or below).

If a patient is withdrawn and experiences adverse events such as

* Admission to hospital
* Amputation
* Ulcer non healing
* Side effects of antibiotics Then details of these events will be subsequently recorded from patient's notes to further complete a health economic evaluation.

Visit 20; Last treatment visit or early termination visit

If the ulcer has not healed after 20 weeks then Visit 20 will be the last treatment visit. Early termination of the study will be carried out if the patient has healed before 20 weeks, or decides to withdraw (and is willing to attend a final visit); or the patient develops a foot ulcer with clinical signs of infection. If the patient has developed side effects from antibiotics and has not taken the antibiotics for more than 72 hours then the patient will be withdrawn from the study.

The unblinded team will always see the patient first.

1. Adverse events will be noted and assessed.
2. Adherence to treatment will be assessed and recorded.
3. Details of the resources that have been used by the patient for treatment of their ulcer will be recorded in order to carry out a health economic evaluation.
4. A physical examination will be carried out.
5. Vital signs will be recorded (body temperature, pulse and blood pressure).
6. Random capillary blood glucose will be measured.
7. Patients with ischaemic ulcers will have their TcPO2 measured.
8. Blood will be collected for the following investigations as per routine clinic practice Calcium and phosphate Renal and liver function Glycated haemoglobin. C- reactive protein Full blood cell count Erythrocyte sedimentation rate Blood glucose Also blood will be taken for high sensitivity C- reactive protein and procalcitonin
9. The patients will be asked to complete Quality of life questionnaire (SF-36) EuroQol-5 questionnaire (EQ-5D)

   Visit procedures by the blinded team
10. Standard ulcer treatment if the ulcer remains unhealed will be carried out. (the removal of callous, any dry skin, any dead tissue in and around the ulcer with a scalpel, ulcer cleansing and application of a dressing)
11. A small tissue sample or ulcer swab will be collected from the ulcer bed for culture and sensitivity
12. Ulcer characteristics (size, depth, site) presence of signs of infection (redness, swelling, pain, malodour, purulent discharge) will be noted.
13. The ulcer circumference will be marked out using sterile graph paper and a marker pen.
14. A digital photograph will be taken of the ulcer.
15. The blinded team will inform the unblinded team whether the ulcer is healed ; if it is not healed whether it is infected or non infected, using the Infectious Disease Society of America/International Working Group on the Diabetic Foot Guidelines (IDSA-IWGDF ) criteria for infection. This will be confirmed by two members of the blinded team

If a patient experiences adverse events such as

* Admission to hospital
* Amputation
* Ulcer non healing
* Side effects of antibiotics Then details of these events will be subsequently recorded from patient's notes, to further complete a health economic evaluation.

Post treatment evaluation

Every patient will be seen 14 days after the last treatment visit or 14 days after the visit when they have been withdrawn from the study. The purpose of this visit is twofold: first to act as a safety visit and secondly, in the case of those patients who had healed at their previous visit to confirm healing.

Visit procedure;

Unblinded team

1. Adverse events will be noted and assessed
2. Body temperature, pulse and blood pressure will be recorded

   Blinded team
3. Standard foot ulcer care will be carried out if the ulcer remains unhealed.
4. If the ulcer had healed at the last visit, then the foot will be examined to confirm healing

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for study participation if he or she meets the following criteria

  * Male or female age 18-85 years inclusive
  * Have been diagnosed with Type 1 or Type 2 diabetes
  * Must be able to speak and understand English and be able to provide meaningful written informed consent .
  * If female, is nonpregnant (negative pregnancy tests at the baseline visit) and nonlactating.
  * If female, is either not of childbearing potential (defined as postmenopausal for ≥ 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy]) or practising one of the following medically-acceptable methods of birth control and agrees to continue with the regimen throughout the duration of the study:

    * Oral, implantable or injectable contraceptives for 3 consecutive months before the baseline visit.
    * Total abstinence from sexual intercourse (≥ 1 complete menstrual cycle before the baseline visit).
    * Intrauterine device
    * Double barrier method (condoms, sponge, diaphragm or vaginal ring with spermicidal jellies or cream)
  * Present with one or more diabetic foot ulcers on or below the malleoli with no clinical signs of infection (using the Infectious Disease Society of America/International Working Group on the Diabetic Foot Guidelines).

Exclusion Criteria:

* Female subjects who are pregnant or breast feeding
* Any known intolerance or allergy or reported adverse reaction to any antibiotics
* Known osteomyelitis
* Patients with foot ulcers with clinical signs of infection
* Ulceration caused primarily by a disease other than diabetes.
* Any other serious disease likely to compromise the outcome of the trial.
* Evidence of critical renal disease (creatinine >300µmol/L)
* Patients taking immunosuppressants or any other preparation which may interfere with healing.
* Participation in another clinical trial in the previous 28 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Time to healing of foot ulceration in each group | 20 weeks

SECONDARY OUTCOMES:
• Percentage of patients who will develop clinical signs of infection over a follow up period of 20 weeks | 20 weeks
• Percentage of patients in each group that are healed at 20 weeks. | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof Mike E Edmonds, FRCP, Principal Investigator — King's College Hospital NHS Trust